CLINICAL TRIAL: NCT04796116
Title: An Exploration of the Role of Metacognition and Masculinity in Men Experiencing Suicidality
Brief Title: Male Suicide and Metacognition
Acronym: MSM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Greater Manchester Mental Health NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Jonothan Orson, Registered Mental Health Nurse, Greater Manchester Mental Health NHS Foundation Trust
Other Study IDs: F485s
Record Dates: First submitted 2021-03-05; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Suicide, Attempted
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Suicide is the act of killing oneself and accounts for one death every 40 seconds around the world. In the UK, over 75% of suicides are completed by men. Suicidal ideation is a symptom of depression and is assessed when diagnosing depressive disorder. Men are three times more likely to complete suicide than women but half as likely to be diagnosed with depression, and therefore risk missing out on potentially lifesaving treatments.

Men experiencing depression and associated suicidality are less likely to demonstrate traditional symptoms such as hopelessness and sadness, and more likely to engage in unhelpful coping strategies such as avoidance through over-working, substance misuse, or risk-taking behaviours, and may feel that they have lost control. Previous research has shown a link between rumination and increased suicidal intent.

Unhelpful coping strategies, distorted beliefs about uncontrollability, and thinking processes such as rumination, are central to the metacognitive model of psychological distress and are targeted in Metacognitive Therapy (MCT).

The aim of this project is to identify if any aspects of the thinking styles described above are present in a sample of men who are suicidal. The project will also explore beliefs about masculinity and how these beliefs might impact help-seeking.

In order to achieve these aims, 15 male service-users without a severe and enduring mental illness, who are receiving care from the Home Based Treatment Team following suicidal thoughts or actions, will be invited to take complete some questionnaires and partake in an interview.

DETAILED DESCRIPTION:
The reduction of suicide is a priority for the Department of Health and Social Care which recommends focusing research and interventions on high-risk groups, such as men. 75% of suicides in the UK are completed by men, it is the biggest killer of men under 45, and 12 men die by suicide each day.

Previous research shows that men may be more likely to mask their symptoms and avoid seeking help from friends, family and professionals. Literature suggests this could be due to the social stigma attached to mental ill health and society's traditional expectations of how men should behave. Evidence also suggests that men may be less likely to present with typical symptoms of depression, such as sadness or hopelessness, and be more likely to engage in activities like overworking, substance misuse, promiscuity and gambling. Studies exploring suicidality in adults have found that increased rumination is linked with higher suicidal intent, and that men in particular may experience accepting antidepressant medication as proof that they have 'lost control'.

Rumination, avoidance, maladaptive coping strategies, and beliefs about uncontrollability are known as 'metacognitions' and are targeted in Metacognitive Therapy (MCT). MCT has a growing evidence base for a range of psychological disorders, including anxiety and depression, and aims to reduce rumination, avoidance, worry, and maladaptive coping strategies, whilst supporting the individual to discover control.

There is a lack of research into how the thinking processes described above present in men who are at risk of suicide. This project aims to contribute to this knowledge base in order to discover whether Metacognitive Therapy (or brief metacognitive interventions) may be a viable treatment option for this population, and worthy of further research. This aim will be achieve by determining which, if any, metacognitions are present in a population of men who are suicidal.

Additionally, the project seeks to explore men's beliefs about masculinity and suicide; and how these beliefs along with the thinking styles previously described, may impact on help-seeking. This could inform future planning of engagement and interventions for this population.

Justification for this research can be found in national reports such as 'The Five Year Forward View' and the 'NHS Long Term Plan', both of which highlight suicide prevention, particularly in high-risk groups such as men, as a priority for clinicians and researchers; more locally, Greater Manchester Mental Health's NHS Foundation Trust's 'Research & Innovation Strategy' commits to conducting research into suicide prevention and improving patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 16+ who are currently receiving care from the Home Based Treatment Team and are experiencing suicidal thoughts and behaviours
* Men with a primary mental health diagnosis of anxiety, depression, acute stress reaction or adjustment disorder, or men with no diagnosis at all
* Men who are able to provide written, informed consent

Exclusion Criteria:

* Women will not be eligible as the aim of this study is to investigate masculinity and its impact on suicidality and help-seeking
* Diagnosis of a severe and enduring mental illness such as Schizophrenia or Bipolar Affective Disorder will be excluded, as their suicidality may be secondary to their diagnosis and more suitable to research within that context
* Non-English-speaking as interviews and assessments will be completed in the English language and are not validated in other languages.
* Unable to provide written, informed consent

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males aged 16+ who are receiving care from the Home Based Treatment Team following suicidal ideation or behaviour and have capacity to provide informed consent to take part.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive Attentional Syndrome Scale (CAS-1) | 2 minutes
  Self-report questionnaire, measuring time spent engaging in metacognitive strategies and conviction in metacognitive beliefs. E.g. First section asks individuals how much time they have spent 'dwelling' on their problems on a scale of 0-8, 0 being none of the time and 8 being all of the time. The latter section asks people to rate beliefs about worry, e.g. 'worrying too much could harm me', on a scale of 0-100 ('0' meaning, 'I do not believe this at all' and '100' meaning, 'I am completely convinced this is true'. There is no 'better' or 'worse' outcome, measure is simply used to describe the population of participants and any common features of the sample.
Metacognitions Questionnaire - 30 (MCQ-30) | 5 minutes
  A self-report questionnaire designed to measure an individual's metacognitive beliefs. The individual rates their agreement with statements such as, 'my worrying is dangerous for me', on a scale of 1-4, 1 meaning 'do not agree' and 4 meaning, 'agree very much'. There is no 'better' or 'worse' outcome, measure is simply used to describe the population of participants and any common features of the sample.
Cognitions Concerning Suicide Scale (CCSS) | 5 minutes
  Self-report questionnaire, where individuals rate how much they agree with beliefs about suicide, such as, 'everyone has the right to commit suicide'; individuals tick whether they 'strongly disagree, disagree, neutral, agree, or strongly agree'. There is no 'better' or 'worse' outcome, measure is simply used to describe the population of participants and any common features of the sample.
Masculine Behaviour Scale (MBS) | 1 minute
  Self-report questionnaire exploring beliefs about masculinity. Individuals rate their agreement with statements about masculinity, such as, 'I don't usually discuss my feelings or emotions with others' by ticking, 'agree, slightly agree, neither agree nor disagree, slightly disagree, disagree'. There is no 'better' or 'worse' outcome, measure is simply used to describe the population of participants and any common features of the sample.
Qualitative Interview | 45 minutes
  Interview conducted using the Metacognitive Profiling Interview Schedule

CONTACTS AND LOCATIONS:
Overall Officials: Jonothan Orson, MA Nursing, Principal Investigator — Greater Manchester Mental Health NHS Foundation Trust
Locations (1):
- Greater Manchester Mental Health NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared. Records will be accessed by the Principal Investigator and other regulatory bodies only for the purpose of audit or investigation.